CLINICAL TRIAL: NCT03876392
Title: Detection of Bone Marrow Metastases With Magnetic Resonance Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Hui, professor, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI001
Record Dates: First submitted 2019-03-04; First posted 2019-03-15 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Bone Marrow Metastases; Magnetic Resonance Imaging
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- magnetic resonance imaging (Experimental): Detection of bone marrow metastases with magnetic resonance imaging
  Interventions: Diagnostic Test: magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging — Compare bone marrow biopsy with magnetic resonance imaging to detect bone marrow metastases

SUMMARY:
The goal of this clinical trial is to study the value and feasibility of magnetic resonance imaging in detection of bone marrow metastases

DETAILED DESCRIPTION:
The patient was diagnosed as bone metastasis by pathology. CT showed no bone marrow biopsy site metastasis (anterior iliac spine or posterior iliac spine). After functional magnetic resonance examination, bone marrow biopsy was performed. Functional magnetic resonance imaging includes conventional SE sequence, T2W SPAIR, e-THRIVE,DWI,IVIM. With bone marrow biopsy as the gold standard, the sensitivity, specificity and coincidence rate of functional MRI in the diagnosis of bone marrow metastasis were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant tumors (solid tumors or hematological malignancies) were definitely diagnosed by pathology or cytology.
2. patients with bone metastases confirmed by more than two imaging examinations.
3. Age 18-75.
4. ECOG score: 0-2.
5. The expected survival time is more than 3 months.
6. Sign the informed consent.

Exclusion Criteria:

1. Imaging findings suggest that bone metastases are present at the bone marrow puncture site.
2. The patient refused bone marrow puncture.
3. Puncture site with infection.
4. Severe coagulation dysfunction.
5. There are implanted instruments in the body, so magnetic resonance imaging can not be performed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity | through study completion, an average of 1 year
  With bone marrow biopsy as the gold standard, the sensitivity of functional MRI in the diagnosis of bone marrow metastasis
specificity | through study completion, an average of 1 year
  With bone marrow biopsy as the gold standard, the specificity of functional MRI in the diagnosis of bone marrow metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People'S Hospital, Shanghai, Other (Non U.s.), China